CLINICAL TRIAL: NCT01906762
Title: Comparing the Effect of Intravenous Morphine and Injectable Acetaminophen on Renal Colic Patients Presenting to the Emergency Department: A Randomized Controlled Trial
Brief Title: Comparing the Analgesic Effect of Intravenous Acetaminophen and Morphine on Patients With Renal Colic Pain Reffering to the Emergency Department: A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seyed Mehdi Pourafzali (Other)
Responsible Party: Sponsor-Investigator, Seyed Mehdi Pourafzali, Emergency Medicine Specialist, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 389456
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Renal Colic
Keywords: Morphine, Acetaminophen, Renal colic, Emergency treatment
MeSH Terms: conditions — Renal Colic | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetaminophen (Experimental): Specified dosage for Acetaminophen was 15 mg/kg. so based on the patient's weight(averagely 70 kg), about 1gr Acetaminophen (one complete Apotel Ampule) was used.
  Interventions: Drug: Acetaminophen
- Morphine (Experimental): Specified dosage for Morphine was 0.1 mg/kg. so based on the patient's weight(averagely 70 kg), about 7 mg Morphine was used.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Acetaminophen — This protocol prepared by a nurse and labeled as Drug A. Since the rapid injection of Acetaminophen can result in hypotension, therefore based on the Apotel Injection Instruction, it must be infused slowly within 15 minutes.
  Other Names: Apotel
  Arms: Acetaminophen
Drug: Morphine — This protocol was prepared by a nurse and labeled as Drug B. Since the rapid injection of Morphine can result in histamine release, therefore it must be infused slowly within 15 minutes. The nurse, who was in charge of infusing pain reliever, was unaware of the type of injected drug.
  Other Names: Morphine Sulfate
  Arms: Morphine

SUMMARY:
Kidney stone is one of the most common diseases in every human society and also Iran. What is normally used to treat renal colic pain is Intravenous Opioid with a variety of side effects including hypotension, respiratory depression and apnea, nausea and vomiting. Regarding less complications of Intravenous Acetaminophen, we aimed to compare it with Intravenous Morphine in management of renal colic pain.

DETAILED DESCRIPTION:
Kidney stone is one of the common diseases of human society which is demonstrated in the form of renal colic. Evidences indicate that renal colic is one of the mot painful conditions that require urgent pain relief treatment.

Patients suffering from renal colic do not usually recover from pain by using oral pain killers or rectal suppositories. Hence, a considerable percentage of these patients are admitted to the emergency department. A bothering and sharp pain is the most common characteristics of renal colic pain that wakes the patient up in the middle of the night. To achieve more relief, patients somehow take unusual positions such as squatting.

What are normally used as pain relievers in emergency department are Non-steroidal anti-inflammatory drugs (NSAIDs) and intravenous Opioids. However, both of these classes of drugs have many side effects.

Another point in this regard which is worthy to be mentioned is that some patients with renal colic complaint are drug addicted, so we have to administer higher dosage of analgesic drugs. According to the statistics provided by the US National Library website, the prevalence of kidney stones around the world in 2005 has been averagely around 140.1% which is considerable. This issue suggests more attention to the field of prevention and treatment.

According to the statistics of kidney stones incidence in Iran, 2.4 out of every 1000 people suffer from this pathologic condition whereas it differs from 0.5 to 2 in every 1000 ones in other countries.

Intravenous Acetaminophen has been imported to our country and introduced with the brand of Apotel. In this regard, we decided to compare the effect of Intravenous Acetaminophen and Morphine on renal colic pain.

ELIGIBILITY:
Inclusion Criteria:

* aged 15 to 80 years
* weight of 60 to 80 kilograms
* known case of renal colic based on physical examination and Ultrasonography

Exclusion Criteria:

* Addiction
* allergic to Opioids and Acetaminophen
* receiving any types of analgesic drugs within previous 6 hours
* known cases of Kidney transplantation
* Patients with known heart failure
* Patients with known Liver failure
* Patients with known Respiratory failure
* Patients with known Renal failure
* cases of Blindness and physical disabilities not able to communicate

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain | 30 Minutes
  patient's pain was assessed by using a Visual Analog Scale Ruler, that rates the amount of pain from 0 to 10 based on patient's confession. Patient's pain was checked out twice: exactly before receiving the pain reliever, and 30 minutes later.